CLINICAL TRIAL: NCT04010084
Title: Effectiveness of Photobiomodulation in Individuals With Chronic Obstructive Pulmonary Disease - Randomized Clinical Trial
Brief Title: Photobiomodulation in Individuals With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OliverDPOC
Record Dates: First submitted 2019-04-25; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Photobiomodulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: the participant will be randomized through a raffle without knowing which group has the active intervention or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Procedure: Placebo group
- Laser group (Active Comparator)
  Interventions: Radiation: Low level laser therapy

INTERVENTIONS:
Radiation: Low level laser therapy — The irradiation will be applied transcutaneously in the sublingual region (3 points on the left side and 3 points on the right side), irradiated for 30 seconds and the total treatment time will be 3 minutes. The group will receive irradiation with a DMC-branded laser EC device, with combined wavelength (660 and 780 nm), 1J of energy per point and output power of 35 mW. A disposable plastic material covering the application pen will be used for hygiene reasons.
  The treatment will be performed twice weekly for a total of 4 consecutive weeks of treatment, and after completion, the patients will be reassessed of all the complementary tests that have been requested.
  Arms: Laser group
Procedure: Placebo group — The irradiation will be applied transcutaneously in the sublingual region (3 points on the left side and 3 points on the right side), irradiated for 30 seconds and the total treatment time will be 3 minutes. The group will receive placebo (with switched-off) irradiation of the DMC-brand laser therapy EC model, with combined wavelength (660 and 780 nm), 1J of energy per point and output power of 35 mW. A disposable plastic material covering the application pen will be used for hygiene reasons.
  The treatment will be performed twice weekly for a total of 4 consecutive weeks of treatment, and after completion, the patients will be reassessed of all the complementary tests that have been requested.
  Arms: Control group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is among the most common chronic respiratory diseases (CKD). Millions of people of all ages suffer from these diseases. COPD is between the fifth and sixth of the leading causes of death in Brazil. It generates an inflammatory pulmonary response that is softened by non-curative treatments and that present serious side effects. Low intensity laser (LBI) or laser therapy has been used for about 50 years to help the healing process, revealing efficient anti-inflammatory and analgesic responses, as well as experimental models of acute and chronic inflammation. However, little is known about its response in inflammatory lung diseases, especially COPD. Some reports indicate that laser therapy may interfere positively by relieving clinical signs, the onset, and the final symptoms of pulmonary inflammation. The present project aims to study the effects of LBI on Chronic Obstructive Pulmonary Disease in patients with pulmonary processes, determine their mechanisms of action and evaluate its effect on patients' functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes;
* Over 18 years of age;
* With a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) for at least 2 years according to the criteria of the clinically stable Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD), free of disease exacerbation in the last 30 days;
* Performing routine outpatient treatment with a pulmonologist;
* Agreement to participate.

Exclusion Criteria:

* Individuals with other comorbidities, such as: Acute Lung Disease, Congestive Heart Failure, Liver Failure, Pulmonary Thromboembolism, Acute Respiratory Distress Syndrome, Neoplasms, HIV Positive, Immunodeficiency, Blood Disorders, Septicemia or recent major surgery.
* Patients with cystic fibrosis and Kartagner's syndrome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-03 (Estimated)

PRIMARY OUTCOMES:
Measure of functional capacity | 4 weeks
  Walk test: In a flat hallway, it will be delimited by two cones and the patient will be guided to walk from one side to the other. The walking speed will be controlled by a "compact disc" that emits beeps (simple BIP) at regular intervals. The test will be interrupted by exhaustion or when the patient is unable to maintain the proposed speed.

SECONDARY OUTCOMES:
TNF-α, IL-1β, IL-6, IL-8, IL-17, IL-10 e IFN-α | 4 weeks
  Quantification of serum levels of interleukin will be performed using Human IL-10 and THF-alpha ELISA MAX (Biolegend) according to the manufacturer's instructions. Briefly, the plates will be coated with anti-IL-10 or anti-TNF-alpha capture monoclonal antibody for 18 h at 8 ° C, washed and then incubated with the reagent provided by the kit to block non-specific binding and to reduce background. Samples will be added to each well at room temperature for 2 h and after washing, the detection antibody solution will be added. The reactions will be revealed with the Avidin-HRP solution and the absorbance will be read at 450nm. They will be evaluated immediately after the end of treatment.
Spirometry | 4 weeks
  The spirometry test will be performed by a physiotherapist using a spirometer apparatus to perform spirometry before and after 20 minutes of bronchodilator administration. The technical procedures, the criteria of acceptability and reproducibility adopted will be those recommended by the Brazilian Consensus of Spirometry. All patients will perform the maneuvers after bronchodilator (salbutamol 400 μg inhalation). They will be evaluated immediately after the end of treatment.
Quality of life assessment questionnaire | 4 weeks
  Saint George's Respiratory Questionnaire (SGRQ): We apply questions related to daily life activities related to the quality of life of patients with COPD. They will be evaluated immediately after the end of treatment.
  The SGRQ addresses aspects related to three areas:
  symptoms, activity and psychosocial impacts that respiratory disease inflicts on the patient. Each domain has a maximum possible score; the points of each answer are summed and the total is referred to as a percentage of this maximum.